CLINICAL TRIAL: NCT04280575
Title: Symptomatic Trial of Angina Assessment Prior to Revascularization: A Placebo-controlled Experiment on Symptoms in Stable Coronary Artery Disease
Brief Title: Symptomatic Trial of Angina Assessment Prior to Revascularization
Acronym: ORBITA-STAR
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other); Mid and South Essex NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 19HH5060
Record Dates: First submitted 2020-02-13; First posted 2020-02-21 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Coronary Artery Disease; Angina, Stable
MeSH Terms: conditions — Coronary Artery Disease; Angina, Stable | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum troponin samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Percutaneous coronary intervention — Coronary artery stenting for stable angina
  Other Names: PCI

SUMMARY:
The principal objective of this research is to determine whether symptoms, induced by confirmed experimental ischaemia, can help us predict which patients will respond to PCI.

ELIGIBILITY:
Inclusion Criteria:

1. Angina or angina-equivalent symptoms
2. Anatomical evidence of a significant single vessel coronary stenosis on diagnostic coronary angiography indicating ≥ 70% stenosis
3. Referred for percutaneous coronary intervention for treatment of stable angina

Exclusion Criteria:

1. Age younger than 18
2. Age older than 85
3. Recent acute coronary syndrome
4. Multivessel coronary artery disease
5. Previous coronary artery bypass graft surgery
6. Significant left main stem coronary disease
7. Chronic total occlusion in the target vessel
8. Contraindication to percutaneous coronary intervention or drug-eluting stent implantation
9. Contraindication to antiplatelet therapy
10. Contraindication to adenosine infusion
11. Severe valvular disease
12. Severe LV systolic impairment
13. Severe respiratory disease
14. Life expectancy less than 2 years, pregnancy, unable to consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with single-vessel coronary artery disease with symptoms of stable angina
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Placebo controlled similarity score during low pressure balloon occlusion of the coronary artery | 30 Days
  Similarity Score (1-10) (Higher Score = Better Outcome)

SECONDARY OUTCOMES:
Change in angina symptom score | 30 Days
  Fractional Change in Angina Frequency (0-1) (Lower Score = Better Outcome)
Change in treadmill exercise time | 30 Days
Change in treadmill time to chest pain | 30 Days
Angina severity as assessed by Canadian Cardiovascular Society Class | 30 Days
  Canadian Cardiovascular Society Class (0-IV) (Lower Score = Better Outcome)
Physical limitation, angina stability, quality of life, angina frequency, freedom from angina as assessed with the Seattle Angina Questionnaire. | 30 Days
  Seattle Angina Questionnaire, (Lower Score = Better Outcome)
Quality of Life assessed with the EQ-5D-5L questionnaire | 30 Days
  (Lower Score = Better Outcome)
Change in dobutamine stress echocardiography score | 30 Days
  (Lower Score = Better Outcome)
Need for anti-anginal medication introduction and uptitration | 30 Days
Anxiety as assessed by the GAD-7 Score | 30 days
  Generalised anxiety and depression - 7 Score. (Lower Score = Better Outcome)
Depression as assessed by the PHQ-9 Score | 30 days
  Patient Health Questionnaire - 9. (Lower Score = Better Outcome)

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Essex Cardiothoracic Centre, Basildon and Thurrock University Hospitals NHS Trust, Basildon, Essex
  - Imperial College Healthcare NHS Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rajkumar CA, Foley MJ, Ahmed-Jushuf F, Chotai S, Simader FA, Mohsin M, Salih A, Ganesananthan S, Bual N, Petraco R, Nijjer SS, Sen S, Sehmi J, Ruparelia N, Dungu JN, Kabir A, Tang K, Gamma R, Davies JR, Kotecha T, Cole GD, Howard JP, Keeble TR, Clesham GJ, O'Kane PD, Harrell FE Jr, Francis DP, Shun-Shin MJ, Al-Lamee RK. The Role of the Collateral Circulation in Stable Angina: An Invasive Placebo-Controlled Study. Circulation. 2025 Dec 2;152(22):1541-1551. doi: 10.1161/CIRCULATIONAHA.125.074687. Epub 2025 Oct 27. PMID 41144984
- [Derived] Rajkumar CA, Foley MJ, Ahmed-Jushuf F, Simader FA, Mohsin M, Ganesananthan S, Nowbar AN, Chotai S, Sen S, Petraco R, Nijjer SS, Sehmi J, Ruparelia N, Dungu JN, Kabir A, Tang K, Gamma R, Davies JR, Kotecha T, Cole GD, Howard JP, Keeble TR, Clesham G, O'Kane PD, Harrell FE Jr, Francis DP, Shun-Shin MJ, Al-Lamee RK. N-of-1 Trial of Angina Verification Before Percutaneous Coronary Intervention. J Am Coll Cardiol. 2024 Jul 2;84(1):1-12. doi: 10.1016/j.jacc.2024.04.001. Epub 2024 May 14. PMID 38752902